CLINICAL TRIAL: NCT00417105
Title: A Multicentric Observational Study on the Removal of Protein-Bound Uremic Retention Solutes in Nocturnal Hemodialysis: A Cross-Sectional Analysis
Brief Title: Protein-Bound Uremic Retention Solutes in Long Nocturnal Hemodialysis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Pieter Evenepoel, University Hospitals Leuven
Other Study IDs: NHD001
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; dialysis adequacy; chronic kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine, dialysate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: hemodialysis twice weekly 4 hours
  Interventions: Procedure: hemodialysis
- 2: nocturnal dialysis twice weekly 8 hours
  Interventions: Procedure: hemodialysis
- 3: nocturnal hemodialysis, 8 hours every other night
  Interventions: Procedure: hemodialysis
- 4: nocturnal hemodialysis, 8 hours, six times per week
  Interventions: Procedure: hemodialysis

INTERVENTIONS:
Procedure: hemodialysis — group 1: twice weekly, four hours
  Groups: 1
Procedure: hemodialysis — group 2: twice weekly, eight hours
  Groups: 2
Procedure: hemodialysis — group 3: every other day, eight hours
  Groups: 3
Procedure: hemodialysis — group 4: six days a week, eight hours
  Groups: 4

SUMMARY:
Although remarkable progress has been made, chronic kidney disease still poses a major burden on both individual patients, as well as on society as a whole. There is a strong inverse relationship between decreasing renal function, as estimated by glomerular filtration rate, and mortality rate, especially death due to cardiovascular disease. The exact cause(s) remain to be elucidated. Uremic toxins might play an important role.

In the course of decreasing renal function the concentration of numerous intracellular and extracellular compounds vary from the non-uremic state. But still increasing number of uremic retention solutes are being identified. Renal replacement strategies aim to remove potentially harmful substances from the body. Traditionally much attention has been paid to small water-soluble molecules such as urea nitrogen and creatinine. Based on the results of the recent HEMO and ADEMEX studies, increases of small water-soluble solute removal above the level reached with modern dialysis techniques - hemodialysis, peritoneal dialysis (HD, PD) - seem not to be advantageous with regard to patient outcome. These findings may point to the importance of other distinct groups of uremic retention solutes. In view of the data described above, protein-bound solutes might be good candidates.

Several advantages of long duration hemodialysis have been observed, including a better control of blood pressure by decreasing extracellular fluid volume, lowering peripheral vascular resistance and improving endothelium-dependent and -independent vasodilation. A normalization of heart rate variability and improvement of left-ventricular function was noted as well. Furthermore, anemia control has been shown to be easier and several nutritional parameters improved in patients treated with long duration HD. The therapy results in higher small water-soluble solute removal, phosphate removal and greater elimination of larger molecules (e.g. β2-microglobulin).

It seems an appealing question whether a better control of the serum levels of protein-bound solutes can be achieved by long duration (nocturnal) hemodialysis. This might be another advantage of this therapeutic modality, or may even in part explain the better outcome of patients treated this way.

The study compares intermittent hemodialysis with long nocturnal hemodialysis with respect to serum concentrations of several protein bound uremic toxins, as well as solute removal.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Maintenance hemodialysis (> 3 months duration)
* Informed consent

Exclusion Criteria:

* No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Maintenance hemodialysis patients
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
removal of protein-bound retention solutes | 1 dialysis session

CONTACTS AND LOCATIONS:
Overall Officials: Björn KI Meijers, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Pieter Evenepoel, MD, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven; Tom Dejagere, MD, Principal Investigator — Virga Jesse Ziekenhuis; Nigel Toussaint, MD, Principal Investigator — Geelong Hospital
Locations (4):
- Australia (2):
  - Monash Medical Centre, Clayton, Victoria
  - Geelong Hospital, Geelong, Victoria
- Belgium (2):
  - Virga Jesse Ziekenhuis, Hasselt, Limburg
  - Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant

REFERENCES:
- [Background] Bammens B, Evenepoel P, Keuleers H, Verbeke K, Vanrenterghem Y. Free serum concentrations of the protein-bound retention solute p-cresol predict mortality in hemodialysis patients. Kidney Int. 2006 Mar;69(6):1081-7. doi: 10.1038/sj.ki.5000115. PMID 16421516
- [Background] Fagugli RM, De Smet R, Buoncristiani U, Lameire N, Vanholder R. Behavior of non-protein-bound and protein-bound uremic solutes during daily hemodialysis. Am J Kidney Dis. 2002 Aug;40(2):339-47. doi: 10.1053/ajkd.2002.34518. PMID 12148107
- [Background] Pierratos A. Daily nocturnal home hemodialysis. Kidney Int. 2004 May;65(5):1975-86. doi: 10.1111/j.1523-1755.2004.00603.x. No abstract available. PMID 15086951